CLINICAL TRIAL: NCT04591132
Title: Technology-based Analysis of Movement Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 130175
Record Dates: First submitted 2020-05-29; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kinematic analysis (Experimental): each patient with a diagnosis of parkinsonism, ataxia, chorea, dystonia or tremor will be asked to perform some motor tasks routinely used in clinical evaluation wearing inertial sensors.
  Interventions: Device: kinematic analysis

INTERVENTIONS:
Device: kinematic analysis — motor tasks appropriate for each diagnosis will be recorder with wearable inertial sensors

SUMMARY:
Objectives: To generate pilot data to investigate the feasibility and the potential use in clinical practice of technology based objective measures of motor performances in patients affected by different movement disorders. To correlate kinematics findings with demographic and clinical details. Trial design and methods: Participants enrolled in prof. Bhatia's movement disorders clinic, will be classifies according to the main movement disorder, specifically, tremor, parkinsonism, dystonia, chorea, ataxia. In the study visit (one day only), they will undergo a clinical evaluation using the appropriate clinical scales (respectively, Fahn-Tolosa-Marin tremor rating scale, MDS-UPDRS Part III, Toronto Western Spasmodic Torticollis Rating Scale 2, Unified Hungtington Disease Rating scale and Scale for the Assessment and Rating of Ataxia) and a kinematic evaluation, using wearables and an infra-red and LED markers system. Then the protocol is concluded and they will continue the routine clinical follow-up

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of parkinsonism and/or dystonia and/or tremor due to:

  1. idiopatic parkinson's disease
  2. atypical parkinsonism
  3. sporadic or inherited/genetic dystonia
  4. young-onset Parkinson's disease
  5. Ataxia syndrome
  6. Choereic syndrome
  7. Essential tremor
  8. Dystonic tremor
* 18 to 80 years of age
* Willing and able to provide informed consent
* able to walk unassisted

Exclusion Criteria:

* Change in pharmacological therapy in the last 3 months.
* Participated in a clinical drug trial up to 3 months before inclusion into the present study
* Orthopaedical comorbidities affecting gait or posture.
* Cognitive deficit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
gait metrics | up to 6 weeks after enrolment
  gait cycles measures (step length, phase duration, number of steps) practice of technology based objective measures of motor performances in patients affected by different movement disorders, to objectively evaluate the disease burden, the efficacy of therapeutic interventions and having a deeper phenotyping of motor disabilities.
tremor peak frequence | up to 6 weeks after enrolment
  fourier analysis for peak frequence of tremor
neck ROM | up to 6 weeks after enrolment
  range of motion of the neck in x,y and z axis
bradykinesia evaluation | up to 6 weeks after enrolment
  amplitude of repeated limb movements over time

SECONDARY OUTCOMES:
correlation with UPDRS gait Item | up to 6 weeks after enrolment
  correlation of gait metrics with UPDRS gait score included.

IPD SHARING:
Plan to Share IPD: No